CLINICAL TRIAL: NCT05515393
Title: A Multicenter, Randomized, Double-blind, Placebo-parallel Controlled, Dose-exploration Phase Ⅱ Clinical Study to Evaluate the Efficacy and Safety of XY03-EA Tablets in the Treatment of Acute Ischemic Stroke
Brief Title: A Study of XY03-EA Tablets in the Treatment of Acute Ischemic Stroke
Acronym: XY03-EA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XY03AIS2001
Record Dates: First submitted 2022-08-08; First posted 2022-08-25 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- XY03-EA Tablet (300mg group) (Experimental): XY03-EA 150 mg/tablet, 2 tablets，three times a day； XY03-EA Placebo 150 mg/tablet, 2 tablets，three times a day； For 90 days, continuous administration Other Name: low dose
  Interventions: Drug: XY03-EA; Drug: XY03-EA Placebo
- XY03-EA Tablet (600mg group) (Experimental): XY03-EA 150 mg/tablet, 4 tablets ,three times a day, For 90 days, continuous administration Other Name:high dose
  Interventions: Drug: XY03-EA
- XY03-EA Placebo Tablet (Placebo Comparator): XY03-EA Placebo Tablet 150 mg/tablet, 4 tablets,three times a day, For 90 days, continuous administration Other Name: placebo
  Interventions: Drug: XY03-EA Placebo

INTERVENTIONS:
Drug: XY03-EA — The sample size was 420 patients, and 140 patients were treated with XY03-EA 300 mg, 600 mg and placebo respectively. The 300-mg group took two tablets of placebo and two tablets of XY03-EA once, three times a day. The 600-mg group took four tablets of XY03-EA once, three times a day. The placebo group took four tablets of placebo once ,three times a day.
  Arms: XY03-EA Tablet (300mg group); XY03-EA Tablet (600mg group)
Drug: XY03-EA Placebo — XY03-EA Placebo
  Arms: XY03-EA Placebo Tablet; XY03-EA Tablet (300mg group)

SUMMARY:
Overall Design: a multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose-exploration study.

Main outcome: 1.To evaluate the efficacy and safety of XY03-EA tablets in the treatment of acute ischemic stroke.

DETAILED DESCRIPTION:
The population is patient who with acute ischemic stroke within 48 hours of onset (including RT-PA intravenous thrombolytic therapy) . The patients were randomized based on being received rt-PA Intravenous thrombolysis or not. Patients who met the inclusion criteria for the protocol were stratified randomly and assigned in a 1:1:1 ratio to three groups: the XY03-EA 300mg, 600mg two-dose group, and the placebo group. The study was divided into 3 stages: screening stage, treatment stage and follow-up stage. The sample size was 420 patients.

Main outcome: 1.To evaluate the efficacy and safety of XY03-EA tablets in the treatment of acute ischemic stroke.

Secondary outcome:

1. Explore the dose-response relationship of XY03-EA tablets in the treatment of acute ischemic stroke, and provide data support for later clinical study;
2. Explore PK characteristics of XY03-EA and its metabolites in patients with acute ischemic stroke based on population PK analysis method.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old (including 18 and 80 years old) ；
2. The patients who diagnosed as acute ischemic stroke according to the Chinese guidelines for the diagnosis and treatment of acute ischemic stroke 2018, total or partial anterior circulation infarction according to the Oxfordshire community stroke classification (OCSP) ;
3. For the patients who received standard intravenous thrombolytic therapy, only the patients who received rt-PA standard intravenous thrombolytic therapy within 4.5 hours of onset were enrolled；
4. Before randomization, 6 points ≤ NIHSS score ≤20 points;
5. From"The last time it seemed normal" to ≤48 hours after the beginning of the study , for the patients who had stroke after waking up or because of aphasia, disturbance of consciousness and other reasons can not accurately time the appearance of symptoms, the time of onset should take the last time the patient showed normally as standard;
6. The patients who first attacked, or the patients who relapsed had a good prognosis after the last attacked , their mRS score was ≤1 before the onset of the disease.
7. Understand and follow the procedure of the study, the patient or guardian agrees to participate, and sign the informed consent form.

Exclusion Criteria:

1. Imaging confirmed intracranial hemorrhagic diseases: hemorrhagic stroke, transformation of symptomatic hemorrhage, epidural hematoma, intracranial hematoma, subarachnoid hemorrhage, intraventricular hemorrhage, traumatic intracerebral hemorrhage, etc.
2. The patients who received urokinase thrombolysis after the onset of the disease were prepared to undergo or had undergone intravascular interventional therapy;
3. Severe disturbance of consciousness:People with consciousness disorder can be defined as "NIHSS score Ia ≥2 points"；
4. Neuroprotective drugs, including Edaravone, Edaravone dexborneol , Butylphthalide, Piracetam and Citicoline, were used after the onset of the disease；
5. Renal insufficiency: serum creatinine > 1.2 times the upper limit of normal, or other known severe renal insufficiency;
6. Liver function damage: AST or ALT > 1.5 times the upper limit of normal value, or other known liver diseases such as acute and chronic hepatitis, cirrhosis, etc.
7. Patients with poor blood pressure control after active treatment: systolic blood pressure ≥220mmHg and/or diastolic blood pressure ≥120mmHg; hypotension: systolic blood pressure ≤80mmHg and/or diastolic blood pressure ≤40mmhg;
8. Severe hyperglycaemia/hypoglycaemia: blood glucose ≥400 mg/dl (22.2 mmol/l) or ≤50 mg/dl (2.8 mmol/L) ;
9. Heart rate less than 50 beats/min and/or heart rate greater than 120 beats/min; Second to third degree atrioventricular block; Patients with previous heart failure (NYHA Class III or IV) , unstable angina, acute myocardial infarction, and severe arrhythmia within 6 months;
10. Patients with dementia, severe Parkinson's disease, mental disorders, claudication, osteoarthropathy, and other disorders that may affect the outcome of treatment；
11. Patients with malignancy, hematologic, digestive, or other serious diseases of the system, or the diseases with bleeding tendency (hemophilia, for example) ；
12. Expected survival time ≤3 months;
13. Patients with a history of severe food or drug allergies, or known allergies to butylphthalide, or celery;
14. Pregnant and lactating or planning pregnancy;
15. Those who had met the criteria for heavy drinking within 3 months before the screening period, that is, daily drinking ≥5 standard drinking quantity (1 standard drinking quantity is equal to 120 ml (2.5 units) of wine, 360 ml (1 can) of beer or 45 ml (1 unit) of liquor) ；
16. Patients with substance abuse or addiction in the past year(narcotic or drugs , for example) ；
17. Those who had taken any clinical trial drug or participated in any drug or device clinical trial or participated in other medical research activities in 3 months before screening and were judged not fit to participate in this study by the investigator;
18. Any other circumstances considered by the investigator might affect the informed consent of the subject or adherence to the study protocol, otherwise the participation of the subject in the study might affect the outcome or his or her own safety.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-09-24 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with Modified Rankin Scale (mRS) score ≤ 1 point at 90 days after administration. | 90 days
  The proportion of patients with Modified Rankin Scale (mRS) score ≤ 1 point at 90 days after administration.
  Modified Rankin Scale, a commonly used scale for measuring the degree of dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. 0 - No symptoms.1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3 - Moderate disability. Requires some help, but able to walk unassisted.4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6 - Dead. The mRS scores between 3 to 6 points are considered to be poor functional outcome.

SECONDARY OUTCOMES:
The proportion of patients with Modified Rankin Scale (mRS) score ≤ 2 point at 14(discharge) , 30,60,90 days after administration. | 14(discharge) , 30,60,90 days
  The proportion of patients with Modified Rankin Scale (mRS) score ≤ 2 point at 14(discharge) , 30,60,90 days after administration;
The proportion of patients with Modified Rankin Scale (mRS) score ≤ 1 point at the 30,60,days after administration; | 30 and 60 days
  The proportion of patients with Modified Rankin Scale (mRS) score ≤ 1 point at the 30,60,days after administration;
The change of NIHSS score from baseline at 14(discharge) , 30,60,90 days after administration; | 14(discharge) , 30,60,90 days
  The change of NIHSS score from baseline at 14(discharge) , 30,60,90 days after administration; The NIHSS is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
The proportion of patients with NIHSS score ≤1 or decrease ≥4 at 30,60, and 90 days after administration; | 30,60, and 90days
  the proportion of patients with NIHSS score ≤1 or decrease ≥4 at 30,60, and 90 days after administration;
The proportion of patients with a BI ≥95 points at 90 days after administration; | 90 days
  The proportion of patients with a BI ≥95 points at 90 days after administration;The BI Scale is a 10-item scale that assesses the ability of daily living. Each item is given 15,10,5 or 0 points depending on whether or not the patient needs help and the degree of help and the time . The total score is 0 to 100 points, the higher the score, the better the independence and self-rationality. According to the assessment results, the ability of daily activities was divided into 3 grades: good, moderate and poor, with a score of more than 60 being good, and basic daily life being self-care; less than or equal to 40 points for poor, most of daily life relying on family care.
The change in MMSE score compared with baseline at 90 days after administration; | 90 days
  The change in MMSE score compared with baseline at 90 days after administration; Mini-mental state examination (MMSE) can comprehensively, accurately and rapidly reflect the intelligence status and the degree of cognitive impairment of the subjects. The scale includes the following 7 aspects: time orientation, place orientation, immediate memory, attention and numeracy, delayed memory, language, visuospatial. The total score of the scale ranged from 0 to 30. The test scores are closely related to the educational level.
New vascular events The proportion of patients with new vascular events | 90 days
  The proportion of patients with new vascular events (ischemic stroke/hemorrhagic stroke/TIA/myocardial infarction/vascular death) within 90 days after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Shijiazhuang Yiling Pharmaceutical Co.,Ltd, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No